CLINICAL TRIAL: NCT07001072
Title: Mitigating Freezing of Gait (FoG) in Parkinson's Disease With Spatiotemporal Haptic Feedback Delivered by Smartshoes
Brief Title: Smartshoes for Freezing of Gait in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Hengameh Zahed, Clinical Assistant Professor of Neurology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 79809
Record Dates: First submitted 2025-05-20; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: freezing of gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Parkinson's disease with freezing episodes (Experimental): Participants perform 3 walking tasks in random order: 1 with receiving vibrotactile feedback in swing-phase of gait, 1 with receiving vibrotactile feedback in metronome (regularly timed) vibration (set at low/medium/fast based on preferred/natural walking speed of the patient at baseline), and another with no vibration.
  Interventions: Device: Smartshoes with haptic vibration feedback
- Parkinson's disease without freezing episodes (Experimental): Participants perform 3 walking tasks in random order: 1 with receiving vibrotactile feedback in swing-phase of gait, 1 with receiving vibrotactile feedback in metronome (regularly timed) vibration (set at low/medium/fast based on preferred/natural walking speed of the patient at baseline), and another with no vibration.
  Interventions: Device: Smartshoes with haptic vibration feedback
- Healthy Controls (Experimental): Participants perform 3 walking tasks in random order: 1 with receiving vibrotactile feedback in swing-phase of gait, 1 with receiving vibrotactile feedback in metronome (regularly timed) vibration (set at low/medium/fast based on preferred/natural walking speed of the patient at baseline), and another with no vibration.
  Interventions: Device: Smartshoes with haptic vibration feedback

INTERVENTIONS:
Device: Smartshoes with haptic vibration feedback — wearable smartshoe with capability‬ to deliver haptic/vibration feedback to assess effect on freezing of gait
  Other Names: NUSHU research

SUMMARY:
This is a pilot research study aimed at evaluating whether an FDA listed wearable shoe with capability to deliver vibration feedback can be safe and tolerable for patients with Parkinson disease and control participants and explore whether such a feedback can be useful for treating freezing of gait (FOG) in patients with Parkinson disease.

ELIGIBILITY:
Inclusion Criteria:

For patients with Parkinson disease:

* diagnosis of PD according to the UK Brain Bank criteria
* Hoehn and Yahr stages 2 to 3 during the ON phase of PD medication
* Self-report episodes of FoG based on item 1 of the NFOG-Q, and score of 3 on item 2, part II

For patients with Parkinson disease withOUT freezing of gait:

* diagnosis of PD according to the UK Brain Bank criteria
* Hoehn and Yahr stages 2 to 3 during the ON phase of PD medication

For all participants (PD with or without freezing, or age-matched controls):

* adult age 40-80
* able to walk 10 minutes at baseline
* able to provide consent
* able to read and write in English at an 8th grade level.

Exclusion Criteria:

For all participants (PD with or without freezing, or age-matched controls)

* moderate to severe peripheral neuropathy (based on self report or clinical exam using vibration tuning fork) which may limit ability to sense the vibratory feedback
* use of orthotics incompatible with the haptic wearable shoes
* severe balance deficits or daily falls at baseline
* patients with dementia (MoCA<18) who are not able to appropriately provide consent for the study
* pregnant persons

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Participant device tolerance survey score | immediately after completion of walking tasks on day 1
Total duration of freezing episodes | Baseline, and day 1 during each walking task (2 min per assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Hengameh Zahed, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No